CLINICAL TRIAL: NCT02788448
Title: Clinical Investigation Plan (CIP) for Safety and Performance Study of Large Hole Vascular Closure Device - FRONTIER III Study
Brief Title: Safety and Performance Study of Large Hole Vascular Closure Device
Acronym: Frontier-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P384-00
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: 18 to 24 F Percutaneous Femoral Arteriotomy Closure
Keywords: Percutaneous vascular closure device; Large hole closure device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VIVASURE CLOSURE DEVICE (Experimental): Large hole closure device
  Interventions: Device: VIVASURE CLOSURE DEVICE

INTERVENTIONS:
Device: VIVASURE CLOSURE DEVICE — Large hole closure device
  Other Names: DP2-FA1-2

SUMMARY:
The purpose of this Clinical Investigation is to validate that the clinical use of the VIVASURE CLOSURE DEVICE™ is safe for the operator, patient and third parties, and to confirm its performance to percutaneously close femoral arterial puncture sites in the range of 18-24 F, post endovascular procedures.

This is a non-inferiority study based on safety. Safety will be assessed by incidence and severity of major complication rates directly related to the VIVASURE CLOSURE DEVICE up to 3 months from implantation is no worse than those associated with cut-down and sutured close.

DETAILED DESCRIPTION:
This study will be a prospective, multi-centred, non-randomized study to investigate the safety and performance of the VIVASURE CLOSURE DEVICE. The study shall not be blinded prior to, during or post the procedure. All patients undergoing a procedure requiring an arteriotomy in the range of 18 to 24 F, via the common femoral artery will be screened against the inclusion/exclusion criteria. If the patient meets the requirements of the clinical investigation, they shall be invited to participate, provide informed consent and shall subsequently be assigned a subject number.

All subjects shall have an immediately post procedure, 24 hour, 1, 3 and 12 month follow-up assessment. Safety data from the follow-ups will be assessed by the Data Safety Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Each patient, or his or her guardian or legal representative, is willing to give informed consent.
* Clinically indicated for an endovascular procedure involving access through the femoral artery, with an access puncture of 18 - 24 F.
* Females who are not pregnant or lactating and not planning to become pregnant ≤ 12 months. A pregnancy test may be performed to confirm this.

Exclusion Criteria:

* Severe acute non-cardiac systemic disease or terminal illness with a life expectancy of less than one year.
* Evidence of systemic bacterial or cutaneous infection, including groin infection.
* Evidence of MRSA (Methicillin-resistant Staphylococcus aureus) colonisation.
* With arterial access other than the common femoral artery.*
* Patients suffering with definitive or potential coagulopathy or platelet count less than 100,000/µl.
* Patient with a haematocrit of less than 30 %.
* A measured activated clotting time (ACT) of greater than 350 seconds immediately prior to sheath removal.*
* If patients are expected to be continuously treated with anticoagulation therapy post-procedure such that their ACT reading is expected to be elevated above 350 seconds for more than 24 hours after the procedure.
* Evidence of arterial diameter stenosis greater than 20 % within 20 mm of the arteriotomy.*
* Circumferential calcification within 20 mm of the arteriotomy.*
* Use of systemic thrombolytic agents within 24 hours prior to or during the catheterisation procedure which cause the concentration of fibrinogen to be less than 100 mg/dl.
* Patients in which the arteriotomy is less than 18 F or greater than 24 F.*
* Known allergy to any of the materials used in the DP2 Device (Refer to Instructions for Use).
* Currently enrolled in any other investigational clinical study, where the primary endpoint has not yet been achieved.
* Patients judged unsuitable for surgical repair of the access site.
* If puncture site is via a vascular graft.
* If there is any indication that the puncture has been made in the profunda femoris or located less than 10 mm above the profunda femoris.*
* Patients with a common femoral artery lumen diameter of less than 7 mm.
* Patients that have a lower extremity amputation from the ipsilateral or contralateral limb.
* Patients that have undergone a percutaneous procedure using a non-absorbable vascular closure device (excluding suture mediated) for haemostasis in the ipsilateral leg.
* Patients that have undergone a percutaneous procedure greater than 8 F in the ipsilateral leg, within the previous 90 days.
* Patients that have undergone a percutaneous procedure of 8 F or less using an absorbable intravascular closure device for haemostasis, in the ipsilateral leg, within the previous 90 days.
* Patients that have undergone a percutaneous procedure of 8 F or less using a suture mediated closure device for haemostasis, in the ipsilateral leg, within the previous 30 days.
* Patients that have undergone a percutaneous procedure of 8 F or less using manual/mechanical pressure for haemostasis in the ipsilateral leg, within the previous 30 days.
* Patients with an acute haematoma of any size, arteriovenous fistula or Pseudoaneurysm at the access site.*
* Significant blood loss/transfusion during interventional procedure or within 20 days prior to procedure requiring transfusion of greater than 4 units of blood.*
* Angiographic evidence of arterial laceration, dissection or stenosis within the external iliac or femoral artery before the use of the DP2 Device.*
* Severe claudication, stenosis of the iliac artery > 50% or previous bypass surgery/stent placement in the region of the vascular access.

  * May not be known until after the patient has given informed consent and the procedure has started. In this event, the DP2 Device should not be used and the patient should be considered excluded from the study and intention to treat analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Major vascular complications [Safety] | up to 3 Months
  Incidence of major vascular complications directly related to study Device (as defined by VARC-2)

SECONDARY OUTCOMES:
Minor vascular complications [Safety] | up to 3 Months
  Incidence of minor vascular complications directly related to the study Device (as defined by VARC-2)
Study device technical success rate [Performance] | within 24 hours
  Technical success rate for the study Device (percentage of subjects not requiring alternative therapy to achieve haemostasis)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med Giovanni Torsello, MD, Principal Investigator — St Fraziskus Hospital, Muenster, Germany
Locations (3):
- Germany (3):
  - The Charité - Universitätsmedizin, Berlin
  - University Hospital Leipzig, Leipzig
  - St Franziskus Hospital, Münster